CLINICAL TRIAL: NCT07298265
Title: Comparison of a Physician-Based Versus Questionnaire-Based Approach to Identify Patients With a High Probability of Psoriatic Arthritis Among Patients With Psoriasis: A Prospective Multicenter Study
Brief Title: Physician- vs Questionnaire-Based Screening for Psoriatic Arthritis in Psoriasis
Acronym: COMPOSITION
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Denis Poddubnyy, Professor, Charite University, Berlin, Germany
Other Study IDs: COMPOSITION2024
Record Dates: First submitted 2025-12-02; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis (PsO); Psoriatic Arthritis (PsA)
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PsO presenting to dermatology, never previously assessed by a rheumatologist for PsA.: Patients with PsO presenting to a dermatologist without a diagnosis of PsA who have not been evaluated for the presence of PsA by a rheumatologist in the past.However, patients with psoriasis who have had an evaluation for the presence of PsA in the past but presenting now with new musculoskeletal symptoms will be eligible.

SUMMARY:
Early diagnosis of psoriatic arthritis (PsA) requires close collaboration between dermatologists (as the skin manifestations of psoriatic disease in most cases precede the musculoskeletal manifestations) and rheumatologists (who are usually responsible for the final diagnosis of PsA and treatment of the musculoskeletal manifestations). Previous epidemiological studies suggest that there may still be a significant proportion of undiagnosed PsA patients among those with psoriasis seen by a dermatologist. At the same time, a diagnostic delay of more than 6 months contributes to poor radiological and functional outcomes in PsA patients. Several screening tools / questionnaires (including the Psoriatic Arthritis Screening Evaluation - PASE, the Toronto Psoriatic Arthritis Screen - ToPAS and its further development - TOPAS 2, the Psoriasis Epidemiology Screening Tool - PEST, and the Early Psoriatic Arthritis Screening Questionnaire - EARP) have been developed and validated in the past decades - all relying mostly on symptoms reported by a patient with psoriasis without an evaluation / confirmation of the presence of musculoskeletal symptoms by a dermatologist. The CONTEST study, which compared three screening tools (PASE, ToPAS and PEST) in a secondary care setting, determined that they all had a good probability of detecting PsA (sensitivity of approximately 80%) but had poor specificity (approximately 35%). Further analysis of the results of the above study has identified the most discriminative questions from each of the three questionnaires, including questions about the back and neck, and these items have been combined to create a new single 8-item screening questionnaire (CONTEST). However, a subsequent study demonstrated a similar performance for the CONTEST and the PEST tools. This poor specificity means that screening questionnaires are often not used in practice and raises a risk of overwhelming rheumatology referrals. In a recent survey of GRAPPA members, most of the participants (consisting of dermatologists, rheumatologists, and patient research partners), suggested that a basic evaluation of MSK symptoms by a dermatologist in addition to the patient-reported symptoms (questionnaire) should be part of the screening / referral process. We hypothesize, therefore, that adding a MSK evaluation by dermatologist in the screening process will be able to improve the outcome of the screening and referral process in relation to the PsA detection. In this study, we plan to evaluate the performance of a physician (dermatologist)-based screening and referral strategy as compared to the strategy based on a questionnaire completed by a patient for the detection of patients with a high probability of a diagnosis of PsA among patients with psoriasis. The primary endpoint will be the proportion of patients diagnosed with PsA among patients with psoriasis referred to a rheumatologist. This will be evaluated in the following groups: 1) PEST-positive and dermatologist-negative patients 2) PEST-positive and dermatologist-positive patients 3) PEST-negative and dermatologist-positive patients 4) PEST-negative and dermatologist-negative patients The primary comparison of the proportions of patients diagnosed with PsA (Fisher's exact test) will be done between the dermatologist-negative vs. positive patients among PEST-positive ones (group 1 vs. group 2).

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Definite diagnosis of psoriasis.
3. Written informed consent.

Exclusion Criteria:

1. Unable or unwilling to give informed consent or to comply with the protocol.
2. Previously assessed by a rheumatologist for the presence of PsA, unless new musculoskeletal symptoms have emerged subsequent to the prior evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis presenting to a dermatologist without a diagnosis of PsA who have not been evaluated for the presence of PsA by a rheumatologist in the past. However, patients with psoriasis who have had an evaluation for the presence of PsA in the past but presenting now with new musculoskeletal symptoms will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Diagnosed with PsA by a Rheumatologist | The study is cross-sectional. Ideally, patients should be seen by both dermatologists and rheumatologists on the same day. However, a window of up to 4 weeks between the dermatology and rheumatology examinations is acceptable.
  The primary outcome will be the proportion of patients diagnosed with PsA by a rheumatologist. This outcome will be evaluated in the following groups:
  1. PEST-positive and dermatologist-negative patients
  2. PEST-positive and dermatologist-positive patients
  3. PEST-negative and dermatologist-positive patients
  4. PEST-negative and dermatologist-negative patients
The proportion of patients diagnosed with PsA. | Cross-sectional assessment with outcome evaluation on the same day or within 28 days
  The primary outcome will be the proportion of patients diagnosed with PsA by a rheumatologist.
  This outcome will be evaluated in the following groups:
  1. PEST-positive and dermatologist-negative patients
  2. PEST-positive and dermatologist-positive patients
  3. PEST-negative and dermatologist-positive patients
  4. PEST-negative and dermatologist-negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network / University Of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided